CLINICAL TRIAL: NCT06209710
Title: Comparing Effectiveness of Balloon Pulmonary Angioplasty Alone vs. Combined With Pulmonary Artery Denervation in Chronic Thromboembolic Pulmonary Hypertension Patients Receiving Standard Medical Therapy
Brief Title: Balloon Pulmonary Angioplasty vs. Combined Approach With Pulmonary Artery Denervation in CTEPH: Effectiveness Comparison
Acronym: BPA-PADN
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boris Dzudovic (Other)
Collaborators: Military Medical Academy, Belgrade, Serbia (Other); Galen Research (Unknown)
Responsible Party: Sponsor-Investigator, Boris Dzudovic, Dr. Boris Dzudovic, MD, PhD, Teaching Assistant at Medical School, University of Defense, Military Medical Academy, Belgrade, Serbia
Organization: Military Medical Academy, Belgrade, Serbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65/2023
Record Dates: First submitted 2024-01-04; First posted 2024-01-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Balloon pulmonary angioplasty; Pulmonary artery denervation; CTEPH

STUDY DESIGN:
Intervention Model Description: Intervention Group: Patients assigned to this group undergo a combination of Balloon Pulmonary Angioplasty (BPA) and Pulmonary Artery Denervation (PADN) alongside standard drug therapy.
  Control Group: Patients in this group receive Balloon Pulmonary Angioplasty (BPA), Sham Pulmonary Denervation and standard drug therapy.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm: BPA + PADN + Standard Drug Therapy (Experimental): Participants in this arm will undergo the combination of Balloon Pulmonary Angioplasty (BPA) and Pulmonary Artery Denervation (PADN) procedures.
  Interventions: Procedure: Balloon Pulmonary Angioplasty combined with Pulmonary Artery Denervation
- Control Arm: BPA + Sham PADN + Standard Drug Therapy (Sham Comparator): Participants in this arm will receive the combination of Balloon Pulmonary Angioplasty (BPA) and standard drug therapy as the control group. Similar to the intervention arm, a denervation catheter will be placed in the same anatomical position, but no further denervation intervention will be performed.
  Interventions: Procedure: Balloon Pulmonary Angioplasty with Sham Pulmonary Artery Denervation

INTERVENTIONS:
Procedure: Balloon Pulmonary Angioplasty combined with Pulmonary Artery Denervation — Participants in the intervention arm will undergo a combination of Balloon Pulmonary Angioplasty (BPA) and Pulmonary Artery Denervation (PADN), as part of this phase 2/3 clinical trial. The trial aims to determine the optimal number of radiofrequency (RF) ablation points required for effective PADN based on pulmonary artery size or diameter. The BPA procedure addresses segmental and subsegmental thrombi masses through pulmonary artery dilation, while the PADN procedure involves the placement of a denervation catheter near the bifurcation of the main pulmonary artery. RF energy is selectively applied, and ablation points are determined based on individual patient characteristics and expected therapeutic effects. This unique approach seeks to customize the intervention to the patient's specific pulmonary anatomy, contributing to the overall effectiveness of the treatment strategy.
  Arms: Intervention Arm: BPA + PADN + Standard Drug Therapy
Procedure: Balloon Pulmonary Angioplasty with Sham Pulmonary Artery Denervation — Participants receive Balloon Pulmonary Angioplasty (BPA) combined with a sham Pulmonary Artery Denervation (PADN) procedure. The sham PADN involves catheter placement mimicking the actual procedure without the application of radiofrequency energy
  Arms: Control Arm: BPA + Sham PADN + Standard Drug Therapy

SUMMARY:
This clinical trial investigates new treatment approaches for chronic thromboembolic pulmonary hypertension (CTEPH), a condition affecting the lungs' blood vessels. CTEPH often develops after repeated blood clots in the lungs, leading to increased pressure and strain on the heart. The study aims to assess the effectiveness of combining two treatments, balloon pulmonary angioplasty (BPA) and pulmonary artery denervation (PADN), in reducing blood pressure in the lungs compared to the standard treatment. Additionally, the trial will explore the impact of these treatments on patients' quality of life. The hope is to improve outcomes and provide valuable insights into managing this challenging condition.

DETAILED DESCRIPTION:
This clinical trial focuses on advancing our understanding and treatment of chronic thromboembolic pulmonary hypertension (CTEPH). CTEPH arises when blood clots in the lungs fail to fully dissolve, leading to the formation of fibrous masses that obstruct blood vessels, increase pulmonary blood pressure, and strain the heart's right ventricle.

The study's primary objective is to evaluate the combined use of two innovative treatments, Balloon Pulmonary Angioplasty (BPA) and Pulmonary Artery Denervation (PADN), in comparison to the standard treatment for CTEPH. BPA involves using a balloon to open narrowed or blocked pulmonary arteries, while PADN is a novel therapy targeting nerve clusters near the main pulmonary artery to reduce blood pressure.

The trial also aims to assess the impact of these treatments on patients' quality of life and clinical improvement measured through the 6-Minute Walk Test Distance (6-MWTD) and the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) questionnaires.In addition to evaluating the combined efficacy of BPA and PADN compared to standard treatment, this clinical trial has a specific objective to customize the PADN intervention based on individual patient characteristics. The study aims to determine the optimal number of radiofrequency (RF) ablation points required for effective PADN, considering the pulmonary artery size or diameter. This innovative approach seeks to tailor the intervention to the unique anatomical features of each patient, enhancing the precision and effectiveness of the treatment strategy.

The study design is a randomized parallel cohort study involving patients with CTEPH in phases 2/3. Patients are divided into two groups-intervention and control-and receive distinct treatment protocols. The intervention group undergoes a combination of BPA, PADN, and standard drug therapy, while the control group receives BPA, sham PADN intervention and standard drug therapy.

The BPA procedure involves accessing the pulmonary artery through the right femoral vein, measuring pressures, and selectively dilating stenosed or occluded branches. After the BPA procedure, PADN is performed by applying radiofrequency energy near the bifurcation of the main pulmonary artery.The sham PADN involves catheter placement mimicking the actual procedure without the application of radiofrequency energy.

The study includes detailed criteria for patient inclusion and exclusion, and patients are closely monitored through scheduled face-to-face visits. The trial plans to enroll approximately 20 patients.

Data management ensures the confidentiality of patient information, and analysis includes a descriptive approach and comparison of mPAP reduction after three months.

The study follows ethical guidelines, Good Clinical Practice, and recommendations from the European Association of Cardiology. Informed consent is a crucial aspect, and patient safety is paramount throughout the trial.

The trial's ultimate goal is to contribute valuable insights into the efficacy of combining BPA and PADN as a potential treatment strategy for CTEPH, aiming to improve patient outcomes and enhance our approach to managing this complex condition.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age 18 - 80 years.
* Diagnosis of chronic thromboembolic heart disease.
* Mean pulmonary arterial pressure (mPAP) >20 mmHg.
* Pulmonary vascular resistance >3 Wood units.
* Presence of organized thrombus masses.
* World Health Organization (WHO) functional class II to IV.

Exclusion Criteria:

* Proximal organized thrombotic masses not suitable for Balloon Pulmonary Angioplasty (BPA) and Pulmonary Artery Denervation (PADN).
* WHO functional class I

Additionally, participants can be excluded from the trial under the following circumstances:

* Withdrawal of consent at any time.
* Failure to complete the treatment as per protocols.
* Protocol violations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean Pulmonary Arterial Pressure (mPAP) | 3 months
  Measure the change in mPAP from baseline to 3 months post-intervention to assess the effectiveness of the combined BPA and PADN therapy.

SECONDARY OUTCOMES:
Quality of Life Assessment | 3 months, and 1 year
  Measure: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) Questionnaire.
  Scale: Units on a scale.
  Scale Details: CAMPHOR consists of three sections:
  Symptoms (Impairment) Scale (0-25): Higher scores indicate a greater extent of symptoms experienced by the patient.
  Activities (Disability) Scale (0-30): Higher scores indicate more significant limitations in performing daily activities affected by chronic thromboembolic pulmonary hypertension.
  Quality of Life Scale (0-25): Higher scores reflect a greater impact of the condition on various aspects of the patient's overall quality of life.
Physical Functionality Assessment | 3 months, and 1 year
  Measure: 6-Minute Walk Test Distance (6-MWTD). Unit of Measure: Meters. Description: The 6-Minute Walk Test evaluates the physical functional capacity of patients with CTEPH. It measures the total distance covered by patients in a six-minute period, providing insight into their exercise tolerance and overall physical performance.
Hemodynamic Response Assessment | 1 year
  Measure: Mean Pulmonary Arterial Pressure (mPAP) change. Unit of Measure: mmHg. Description: Assesses mPAP reduction after 1 year
Adverse Events | 3 months, abd 1 year
  Measure: Number of Participants with Documented and Categorized Adverse Events, Including Intensity and Type (e.g., cardiovascular events, bleeding events, procedural complications), to Evaluate Safety.
Survival Rates | 1 year
  Monitor one-year survival rate to provide insights into the long-term outcomes of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Obradovic, MD, PhD, Principal Investigator — Clinic of Cardiology, Military Medical Academy, Belgrade, Serbia
Locations (1):
- Military Medical Academy, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
We intend to share de-identified individual participant data, excluding any personally identifiable information (PII), to protect participant privacy.
  Data sharing is planned to commence after the completion of the trial and the release of the main study results. The exact timing for data sharing will be in compliance with regulatory requirements and ethical considerations.
  Access to the shared data will be granted to researchers who submit formal requests outlining their research objectives, methodologies, and plans for data usage. A data sharing agreement will be established to ensure adherence to ethical standards and protection of participant confidentiality.
  Data will be shared in a standardized and machine-readable format, allowing for compatibility with various statistical analysis tools and software.
  The study team is committed to providing necessary documentation and support to facilitate the appropriate use and interpretation of the shared data.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data sharing is planned to commence after the completion of the trial and the release of the main study results. The exact timing for data sharing will be in compliance with regulatory requirements and ethical considerations.
Access Criteria: Access to the shared data will be granted to researchers who submit formal requests outlining their research objectives, methodologies, and plans for data usage. A data sharing agreement will be established to ensure adherence to ethical standards and protection of participant confidentiality.

REFERENCES:
- [Background] Chen SL, Zhang FF, Xu J, Xie DJ, Zhou L, Nguyen T, Stone GW. Pulmonary artery denervation to treat pulmonary arterial hypertension: the single-center, prospective, first-in-man PADN-1 study (first-in-man pulmonary artery denervation for treatment of pulmonary artery hypertension). J Am Coll Cardiol. 2013 Sep 17;62(12):1092-1100. doi: 10.1016/j.jacc.2013.05.075. Epub 2013 Jul 10. PMID 23850902
- [Background] Zhang H, Wei Y, Zhang C, Yang Z, Kan J, Gu H, Fan F, Gu H, Wang Q, Xie D, Zhang G, Guo X, Yin Y, Jin B, Zhou H, Yang Z, Wang Z, Xin Y, Zhang C, Meng L, Wang X, Sun J, Zhao C, Zhang J, Yan X, Chen F, Yao C, Stone GW, Chen SL. Pulmonary Artery Denervation for Pulmonary Arterial Hypertension: A Sham-Controlled Randomized PADN-CFDA Trial. JACC Cardiovasc Interv. 2022 Dec 12;15(23):2412-2423. doi: 10.1016/j.jcin.2022.09.013. Epub 2022 Sep 18. PMID 36121246